CLINICAL TRIAL: NCT01886625
Title: Single-port Thoracoscopic Sympathicotomy for Treatment of Complex Regional Pain Syndrome Type I, a Feasibility Study.
Brief Title: Single-port Thoracoscopic Sympathicotomy in Complex Regional Pain Syndrome Type I (CRPS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No local inclusions
Sponsor: University of Groningen (Other)
Responsible Party: Principal Investigator, Michiel Kuijpers, Principal Investigator, University of Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL41466.042.12
Record Dates: First submitted 2013-03-24; First posted 2013-06-26 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Complex Regional Pain Syndrome Type I of the Upper Limb
MeSH Terms: conditions — Reflex Sympathetic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sympathicotomy (Experimental): unilateral single-port VATS sympathicotomy
  Interventions: Procedure: unilateral single-port VATS sympathicotomy

INTERVENTIONS:
Procedure: unilateral single-port VATS sympathicotomy

SUMMARY:
Background of the study: CRPS type-1 is a pain syndrome that usually develops after an initiating noxious event (e.g. fracture) in an extremity. Although treatment options life dimethyl-sulphoxide (DMSO), N-acetylcysteine (NAC) and intensive physical therapy exist, the treatment effect is often unsatisfactory, even leading to amputation of the extremity. Surgical treatment of chronic pain disorders by dividing the sympathetic chain is an established treatment. Its more invasive nature has prevented widespread application. After introduction of minimal invasive techniques in recent years, the UMCG has now devised a truly minimal invasive, yet safe and effective thoracoscopic technique, that requires only a single 1 cm long incision in the anterior axillary line. This technique is developed as treatment for primary focal axillary and palmar hyperhidrosis, and is performed in over 50 patients producing very satisfying results. This fact has led to the hypothesis that this same surgical technique can offer this group of chronic pain patients a safe, effective treatment modality.

Objective of the study: The effect of the intervention on pain an regain of function in de affected extremity. This will be quantified in multiple questionnaires at baseline and three follow-up points, and by clinical evaluation of the hand function at baseline and two follow-up points.

Study design: Single center prospective feasibility study

ELIGIBILITY:
Inclusion Criteria:

Age 18 - 65 years.

* ASA 1 en 2.
* CRPS-1 defined according to IASP-Bruehl criteria at the wrist or lower arm level.

  1. Continuing pain which is disproportionate to any inciting event
  2. Must report at least one symptom in each of the four following categories

     * Sensory: reports of hyperesthesia
     * Vasomotor: reports of temperature asymmetry, skin color change or asymmetry.
     * Sudomotor/edema: reports of edema, sweating changes, sweating asymmetry
     * Motor/trophic: reports of decreased range of motion, motor dysfunction (weakness, tremor, dystonia), trophic changes (hair, nail, skin)
  3. Must display at least one sign in two or more of the following categories:

     * Sensory: evidence of hyperalgesia (to pinprick) and/or allodynia (to light touch)
     * Vasomotor: evidence of temperature asymmetry, color changes, asymmetry
     * Sudomotor/edema: evidence of edema, sweating changes, sweating asymmetry
     * Motor/trophic: evidence of decreased range of motion, motor dysfunction (weakness, tremor, dystonia), trophic changes (hair, nail, skin)

Exclusion Criteria:

Known COPD > Gold class 1.

* History of smoking > 20 pack years, due to higher risk of complications following unilateral lung- deflation and re-insufflation.
* Documented substance addiction.
* Previous intra-thoracic pleural drainage on affected side.
* Previous thoracic surgery on affected side (including sternotomy). - Gross pulmonary or pleural abnormalities on chest X-ray.
* Pregnancy, determined by preoperative pregnancy test.
* Unsuitable anatomy (e.g. due to severe physical malformations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change in perceived pain measured in Visual Analogue Scale | Baseline, 1, 3 and 6 months postoperative

SECONDARY OUTCOMES:
Change in function in extremity | Baseline, 1 and 6 months after intervention
  Strength in fingers, maximal flexion/extension in all digits, volumetric measurement, timing simple daily tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo A Mariani, MD, PhD, Study Chair — University Medical Center Groningen; Michiel Kuijpers, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands